CLINICAL TRIAL: NCT02153476
Title: A Safety And Efficacy Study Of Alg-1001 In Human Subjects With Symptomatic Focal Vitreomacular Adhesion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allegro Ophthalmics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMA-202
Record Dates: First submitted 2014-05-27; First posted 2014-06-03 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Symptomatic Focal Vitreomacular Adhesion
MeSH Terms: interventions — risuteganib; Hanks Balanced Salt Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2.0mg of ALG-1001 (Experimental): 2.0mg of ALG-1001
  Interventions: Drug: 2.0mg of ALG-1001
- Intravitreal injection in 0.05cc balanced salt solution. (Placebo Comparator): Balanced Salt Solution
  Interventions: Drug: Balanced Salt Solution

INTERVENTIONS:
Drug: 2.0mg of ALG-1001
  Arms: 2.0mg of ALG-1001
Drug: Balanced Salt Solution
  Arms: Intravitreal injection in 0.05cc balanced salt solution.

SUMMARY:
Evaluate the safety and efficacy of ophthalmic intravitreal injection of ALG-1001 in human subjects with symptomatic focal vitreomacular adhesion

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic focal vitreomacular adhesion
2. Vitreomacular traction syndrome
3. Stage 1 and 2 macular holes, ≤ 350 µm
4. BCVA of 20/25 Early Treatment Diabetic Retinopathy Study (ETDRS) or worse in the study eye
5. BCVA of 20/800 ETDRS or better in the fellow eye
6. Male or female subjects, 18 years of age or older
7. Signed Informed Consent

Exclusion Criteria:

1. High myopes > -8.0 D spherical equivalent
2. History of prior vitrectomy in the study eye
3. History of photocoagulation to the retina in the study eye
4. Macular hole in the study eye > 350 µm
5. Subjects with epiretinal membranes in the study eye
6. Subjects with broad VMA, defined as VMA of >1500 µm
7. Subjects with proliferative Diabetic Retinopathy (DR), neovascular Age-related Macular Degeneration (AMD), or retinal vascular occlusion in the study eye
8. Subjects with aphakia in the study eye
9. Subjects with uncontrolled glaucoma
10. Subjects with lenticular or zonular instability
11. Subjects with prior ocular surgery or intravitreal injection in the study eye within 90 days of study enrollment
12. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - California Retina Consultants, Santa Barbara, California
  - Center for Retinal and Macular Disease, Winter Haven, Florida
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravitreal Injection in 0.05cc BSS: Balanced Salt Solution
  Balanced Salt Solution
Period: Overall Study
Arm/Group | 2.0mg of ALG-1001 | Intravitreal Injection in 0.05cc BSS
Started | 23 | 22
Completed | 22 | 22
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.0mg of ALG-1001 | Intravitreal Injection in 0.05cc BSS | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 39
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Full Range); unit: years] | 49 [25 to 70] | 49 [25 to 70] | 49 [25 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 12 | 12 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Release of Vitreo Macular Adhesion (VMA) by Optical Coherence Tomography (OCT)
Description: The primary endpoint of this study is observation of pharmacologic resolution of VMA, with VMA defined as vitreous adhesion to the macula within a 6mm central retinal field surrounded by elevation of the posterior vitreous cortex as seen on OCT.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | 2.0mg of ALG-1001 | Intravitreal Injection in 0.05cc BSS
Number analyzed (Participants) | 23 | 22
Participants | 4 | 0

ADVERSE EVENTS:
Arm/Group | 2.0mg of ALG-1001 | Intravitreal Injection in 0.05cc BSS
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No